CLINICAL TRIAL: NCT03821727
Title: Outcome of Hematopoietic Stem Cell Transplantation in Philadelphia Positive Acute Lymphoblastic Leukemia in the Era of Tyrosine Kinase Inhibitors. A Registry-based Study of the Italian Blood and Marrow Transplantation Society (GITMO)
Brief Title: SCT in Ph Positive Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: CANDONI ANNA (Other)
Collaborators: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor-Investigator, CANDONI ANNA, Principal Investigator, Clinical Professor, University Hospital, Udine, Italy
Organization: University Hospital, Udine, Italy (Other)
Other Study IDs: PRN°0068937
Record Dates: First submitted 2019-01-19; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Philadelphia Positive Acute Lymphoblastic Leukemia; SCT
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hematopoietic Stem Cell Transplantation — Hematopoietic Stem Cell Transplantation in Acute Leukemia Ph positive

SUMMARY:
This study includes a registry-based, nationwide analysis to describe the clinical outcome of adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL) who underwent an allogeneic hematopoietic stem cell transplantation (HSCT) after a Tyrosine Kinase Inhibitors (TKI)-based treatment.

DETAILED DESCRIPTION:
This was a retrospective nationwide analysis based on registry data collected by GITMO. Inclusion criteria were: 1) diagnosis of Ph+ ALL; age ≥18 years at transplant; 2) patients receiving first allogeneic HSCT from any donor (HLA-identical sibling donor (MSD), unrelated donor (UD) or alternative donor (haploidentical or cord blood) between 2005 and 2016 in a GITMO center; 3) TKI-based treatment prior to HSCT; 4) patients with available pre-transplant MRD status, as well as complete clinical data and outcome. Data were extracted from the GITMO Registry (PROMISE Registry).

The endpoints of the study were: OS, progression-free survival (PFS), cumulative incidence of relapse (CIR), non-relapse mortality (NRM), cumulative incidence of extensive chronic graft versus host disease (cGVHD), rate of minimal residual disease (MRD) negativity and the rate of complete cytologic remission (CR) before and after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ph+ ALL; age ≥18 years at transplant.
* Patients receiving first allogeneic HSCT from any donor (HLA-identical sibling donor (MSD), unrelated donor (UD) or alternative donor (haploidentical or cord blood) between 2005 and 2016 in a GITMO center.
* TKI-based treatment prior to HSCT.
* Patients with available pre-transplant MRD status, as well as complete clinical data and outcome.

Exclusion Criteria:

* All cases without one or more of inclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data were extracted from the GITMO Registry (PROMISE Registry). All patients received a first allogeneic HSCT from any donor.
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS). | 5 years
  as reported

SECONDARY OUTCOMES:
Rate of complete cytologic remission (CR) before and after transplant. | Baseline and 3 months after SCT
  As reported
Rate of minimal residual disease (MRD). | Baseline and 3 months post SCT
  As reported
Cumulative incidence of extensive chronic graft versus host disease (cGVHD). | 5 years
  as reported

OTHER OUTCOMES:
Progression-free survival (PFS). | 5 years
  as reported
Cumulative incidence of relapse (CIR). | 5 years
  as reported
Non-relapse mortality (NRM). | 5 years
  as reported

CONTACTS AND LOCATIONS:
Overall Officials: Renato Fanin, Professor, Principal Investigator — University of Udine
Locations (2):
- Italy (2):
  - GITMO Centers and GITMO CLINICAL OFFICE-AOU-IRCSS San Martino-Ge, Genova
  - University Hospital, Udine, Udine

IPD SHARING:
Plan to Share IPD: No
Data were extracted from the GITMO Registry (PROMISE Registry). All patients included in the registry signed an informed consent form. The study was conducted in compliance with current national and European legislation on clinical trials, in accordance with the Helsinki Declaration and the principles of good clinical practice (GCP). This study was approved by the GITMO board and by the institutional review board of the coordinating center (Hematology-University of Udine) and from institutional review boards of all participating centers.

REFERENCES:
- [Derived] Candoni A, Rambaldi A, Fanin R, Velardi A, Arcese W, Ciceri F, Lazzarotto D, Lussana F, Olivieri J, Grillo G, Parma M, Bruno B, Sora F, Bernasconi P, Saccardi R, Foa R, Sessa M, Bresciani P, Giglio F, Picardi A, Busca A, Sica S, Perruccio K, Zucchetti E, Diral E, Iori AP, Colombo AA, Tringali S, Santarone S, Irrera G, Mancini S, Zallio F, Malagola M, Albano F, Carella AM, Olivieri A, Tecchio C, Dominietto A, Vacca A, Sorasio R, Orciuolo E, Risitano AM, Leotta S, Cortelezzi A, Mammoliti S, Oldani E, Bonifazi F; GITMO. Outcome of Allogeneic Hematopoietic Stem Cell Transplantation in Adult Patients with Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia in the Era of Tyrosine Kinase Inhibitors: A Registry-Based Study of the Italian Blood and Marrow Transplantation Society (GITMO). Biol Blood Marrow Transplant. 2019 Dec;25(12):2388-2397. doi: 10.1016/j.bbmt.2019.07.037. Epub 2019 Aug 7. PMID 31400502